CLINICAL TRIAL: NCT00589381
Title: Phase I Trial of Fenretinide (4-HPR, NSC 374551) Lym-X-Sorb™ (LXS) Oral Powder (4-HPR/LXS Oral Powder) (4-HPR) in Adults With Solid Tumors and Lymphomas
Brief Title: Fenretinide Lym-X-Sorb™ in Treating Patients With Recurrent or Resistant Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 080030; 08-C-0030; NCI-P07187; CDR0000580777
Record Dates: First submitted 2007-12-20; First posted 2008-01-09 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; recurrent adult Hodgkin lymphoma; recurrent adult T-cell leukemia/lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; Waldenström macroglobulinemia; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent small lymphocytic lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell

INTERVENTIONS:
Drug: fenretinide lipid matrix

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fenretinide Lym-X-Sorb™ , work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I trial is studying the side effects and best dose of fenretinide Lym-X-Sorb™ in treating patients with recurrent or resistant solid tumors or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of fenretinide Lym-X-Sorb™ oral powder (4-HPR/LXS oral powder) in patients with recurrent and/or resistant solid tumors or lymphomas.
* To define the toxicities of 4-HPR/LXS oral powder in these patients.
* To determine the plasma pharmacokinetics of 4-HPR/LXS oral powder in these patients.

Secondary

* To determine the level of fenretinide delivered as 4-HPR/LXS oral powder in normal peripheral blood mononuclear cells.

OUTLINE: This is a multicenter study.

Patients receive oral fenretinide Lym-X-Sorb™ oral powder (4-HPR/LXS oral powder) (mixed in food carriers) three times daily on days 1-7. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease response or better may receive additional courses of treatment at the discretion of the treating physician and principal investigator.

Blood samples are collected periodically for pharmacokinetic and pharmacodynamic studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed (by the NIH pathology department) diagnosis of 1 of the following:

  * Solid tumor malignancy that is metastatic or unresectable
  * Lymphoma for which standard treatment or curative measures do not exist, or are associated with minimal patient survival benefit
* Recurrent and/or resistant disease
* Measurable or evaluable disease
* No known brain metastases

  * Patients whose brain metastatic disease status has remained stable for ≥ 3 months after treatment may be eligible at the discretion of the principal investigator (without steroids or anti-seizure medications)

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy ≥ 3 months
* Absolute neutrophil count ≥ 1,500/µL
* Platelets ≥ 100,000/µL (CTCAE v.3 grade 1 thrombocytopenia allowed if explained by involvement of the bone marrow by lymphoma)
* Total bilirubin ≤ 1.5 times normal institutional limits (2.5 mg/dL for patients with Gilbert's syndrome)
* AST (SGOT)/ALT (SGPT) ≤ 2.5 times upper limit of normal (ULN)
* Creatinine < 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use two methods of birth control, including at least one highly effective method (e.g., intrauterine device [IUD], hormonal birth control pills/injections/implants, tubal ligation or partner's vasectomy), and one additional effective method (e.g., latex condoms, diaphragm, or cervical cap), prior to, during, and for 2 months after completion of study treatment

  * Men must use a latex condom every time they have sexual intercourse during therapy and for 2 months after discontinuing fenretinide, even if they have had a successful vasectomy
* No clinically significant illnesses which could compromise participation in the study, including, but not limited to, any of the following:

  * Active or uncontrolled infection
  * Immune deficiencies or confirmed diagnosis of HIV infection
  * Uncontrolled diabetes
  * Uncontrolled hypertension
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Myocardial infarction within the past 6 months
  * Uncontrolled cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* No known wheat gluten allergy or allergy or sensitivity to the study drug
* No history of pancreatitis as evidenced by elevated amylase or lipase ≥ grade 2 and accompanied by symptoms of pancreatitis (e.g., abdominal pain)

PRIOR CONCURRENT THERAPY:

* Recovered from adverse events and/or toxicity due to prior chemotherapy or biologic therapy
* No chemotherapy or biologic therapy within 4 weeks prior to entering the study (6 weeks for nitrosoureas, mitomycin C, or UCN-01)
* At least 1 month since any prior radiotherapy or major surgery
* At least 2 weeks since any prior administration of study drug in an exploratory IND/phase 0 study
* Patients receiving bisphosphonates for any cancer or undergoing androgen deprivation therapy for prostate cancer are eligible for this therapy
* No concurrent sulfonamides
* No other concurrent investigational agents
* No other concurrent cancer chemotherapy, or immunomodulating agents (including systemic corticosteroids)
* Patients must not take any drugs suspected of causing pseudo tumor cerebri, including any of the following:

  * Tetracycline
  * Nalidixic acid
  * Nitrofurantoin
  * Phenytoin
  * Sulfonamides
  * Lithium
  * Amiodarone
  * Vitamin A (except as part of routine total parenteral nutrition vitamin supplements or in a single daily standard dose oral multivitamin supplement)
* No concurrent herbal supplements or other alternative therapy medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-08; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of 4-HPR/LXS oral powder
Safety
Toxicity

SECONDARY OUTCOMES:
Level of fenretinide in normal peripheral blood mononuclear cells

CONTACTS AND LOCATIONS:
Overall Officials: Shivaani Kummar, MD, Study Chair — NCI - Medical Oncology Branch
Locations (4):
- United States (4):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland

REFERENCES:
- [Result] Kummar S, Gutierrez ME, Maurer BJ, Reynolds CP, Kang M, Singh H, Crandon S, Murgo AJ, Doroshow JH. Phase I trial of fenretinide lym-x-sorb oral powder in adults with solid tumors and lymphomas. Anticancer Res. 2011 Mar;31(3):961-6. PMID 21498721